CLINICAL TRIAL: NCT00067938
Title: Lamictal for Use in Treatment of Bipolar Disorder In Adults. A Practical Clinical Assessment of Tolerability and Clinical Effectiveness.
Brief Title: Bipolar Study in Adults at Least 18 Years of Age
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCA40917
Record Dates: First submitted 2003-09-03; First posted 2003-09-05 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Bipolar Disorder
Keywords: bipolar disorder; lamotrigine
MeSH Terms: conditions — Bipolar Disorder | interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other): Open label single arm study
  Interventions: Drug: lamotrigine

INTERVENTIONS:
Drug: lamotrigine — Lamotrigine

SUMMARY:
Bipolar study of tolerability, clinical response and patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar I disorder.
* Must be on a stable regimen of psychiatric medication for at least 2 months prior to study.
* If female, must not be pregnant, or must be incapable of conceiving or be taking steps to prevent conception.

Exclusion Criteria:

* Patients with a clinically significant psychiatric or physiologic comorbidity including significant substance abuse, depression or mania which is of an unstable of progressive nature that could interfere in participation of this study.
* Presence of untreated thyroid disease.
* Patient is actively suicidal or homicidal.
* Patient has history of severe hepatic or renal insufficiency.
* Patient is currently participating in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2003-08; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the rate of rash during 12 weeks. | 12 Weeks

SECONDARY OUTCOMES:
Change from baseline in Week 5 and Week 12 Clinical Global Impression-Bipolar version (CGI-BP) Severityand Improvement scores. | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (257):
- United States (257):
  - GSK Investigational Site, Albertville, Alabama
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Fairhope, Alabama
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Tuscaloosa, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Rogers, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Fort Smith, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, North Little Rock, Arkansas
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Burbank, California
  - GSK Investigational Site, Campbell, California
  - GSK Investigational Site, Cerritos, California
  - GSK Investigational Site, El Centro, California
  - GSK Investigational Site, Fairfield, California
  - GSK Investigational Site, La Mesa, California
  - GSK Investigational Site, Laguna Hills, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Oceanside, California
  - GSK Investigational Site, Petaluma, California
  - GSK Investigational Site, Poway, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Santa Barbara, California
  - GSK Investigational Site, Sherman Oaks, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, West Hollywood, California
  - GSK Investigational Site, Boulder, Colorado
  - GSK Investigational Site, Fort Collins, Colorado
  - GSK Investigational Site, Hamden, Connecticut
  - GSK Investigational Site, Mansfield Center, Connecticut
  - GSK Investigational Site, Norwich, Connecticut
  - GSK Investigational Site, Wethersfield, Connecticut
  - GSK Investigational Site, Newark, Delaware
  - GSK Investigational Site, Wilmington, Delaware
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Altamonte Springs, Florida
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Boynton Beach, Florida
  - GSK Investigational Site, Bradenton, Florida
  - GSK Investigational Site, Brandon, Florida
  - GSK Investigational Site, Casselberry, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Coral Springs, Florida
  - GSK Investigational Site, Davie, Florida
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, Destin, Florida
  - GSK Investigational Site, Fort Walton Beach, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Jacksonville Beach, Florida
  - GSK Investigational Site, Lakeland, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, North Miami, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Orange City, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Palm Beach Gardens, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Syracuse, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Wilton Manors, Florida
  - GSK Investigational Site, Winter Park, Florida
  - GSK Investigational Site, Zephyrhills, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Roswell, Georgia
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Warner Robins, Georgia
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Alton, Illinois
  - GSK Investigational Site, Bourbonnais, Illinois
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, East Moline, Illinois
  - GSK Investigational Site, Evergreen Park, Illinois
  - GSK Investigational Site, Fairview Heights, Illinois
  - GSK Investigational Site, Granite City, Illinois
  - GSK Investigational Site, Joliet, Illinois
  - GSK Investigational Site, Libertyville, Illinois
  - GSK Investigational Site, Lisle, Illinois
  - GSK Investigational Site, Oakbrook Terrace, Illinois
  - GSK Investigational Site, Orland Park, Illinois
  - GSK Investigational Site, Park Ridge, Illinois
  - GSK Investigational Site, Rockford, Illinois
  - GSK Investigational Site, Schaumburg, Illinois
  - GSK Investigational Site, Vernon Hills, Illinois
  - GSK Investigational Site, Wheaton, Illinois
  - GSK Investigational Site, Danville, Indiana
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Fort Wayne, Indiana
  - GSK Investigational Site, Lafayette, Indiana
  - GSK Investigational Site, Mishawaka, Indiana
  - GSK Investigational Site, Plymouth, Indiana
  - GSK Investigational Site, Valparaiso, Indiana
  - GSK Investigational Site, Cedar Rapids, Iowa
  - GSK Investigational Site, Dubuque, Iowa
  - GSK Investigational Site, Leavenworth, Kansas
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Shawnee Mission, Kansas
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Hopkinsville, Kentucky
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Houma, Louisiana
  - GSK Investigational Site, Lake Charles, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Annapolis, Maryland
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Batlimore, Maryland
  - GSK Investigational Site, Burtonsville, Maryland
  - GSK Investigational Site, Ellicott City, Maryland
  - GSK Investigational Site, Gaithersburg, Maryland
  - GSK Investigational Site, Glen Burnie, Maryland
  - GSK Investigational Site, Laurel, Maryland
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Towson, Maryland
  - GSK Investigational Site, Adrian, Michigan
  - GSK Investigational Site, Bay City, Michigan
  - GSK Investigational Site, Benton Harbor, Michigan
  - GSK Investigational Site, Bloomfield Hills, Michigan
  - GSK Investigational Site, Brownstown Township, Michigan
  - GSK Investigational Site, Clinton Township, Michigan
  - GSK Investigational Site, East Lansing, Michigan
  - GSK Investigational Site, Farmington Hills, Michigan
  - GSK Investigational Site, Flint, Michigan
  - GSK Investigational Site, Mount Clemens, Michigan
  - GSK Investigational Site, Rochester Hills, Michigan
  - GSK Investigational Site, Royal Oak, Michigan
  - GSK Investigational Site, Duluth, Minnesota
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Oakdale, Minnesota
  - GSK Investigational Site, Flowood, Mississippi
  - GSK Investigational Site, Gulfport, Mississippi
  - GSK Investigational Site, Joplin, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Billings, Montana
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Manchester, New Hampshire
  - GSK Investigational Site, Long Branch, New Jersey
  - GSK Investigational Site, Princeton, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Las Cruces, New Mexico
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Amityville, New York
  - GSK Investigational Site, Farmingdale, New York
  - GSK Investigational Site, Latham, New York
  - GSK Investigational Site, New Rochelle, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Olean, New York
  - GSK Investigational Site, Port Jefferson, New York
  - GSK Investigational Site, Smithtown, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Cary, North Carolina
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Cornelius, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Fayetteville, North Carolina
  - GSK Investigational Site, Forest City, North Carolina
  - GSK Investigational Site, Goldsboro, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, High Point, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Avon Lake, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cuyahoga Falls, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Warren, Ohio
  - GSK Investigational Site, Youngstown, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Milwaukie, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Colmar, Pennsylvania
  - GSK Investigational Site, Doyletown, Pennsylvania
  - GSK Investigational Site, Kingston, Pennsylvania
  - GSK Investigational Site, McKeesport, Pennsylvania
  - GSK Investigational Site, Media, Pennsylvania
  - GSK Investigational Site, Natrona Heights, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Reading, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Moncks Corner, South Carolina
  - GSK Investigational Site, North Charleston, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Cordova, Tennessee
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Madison, Tennessee
  - GSK Investigational Site, Murfreesboro, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Bedford, Texas
  - GSK Investigational Site, Conroe, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Humble, Texas
  - GSK Investigational Site, Irving, Texas
  - GSK Investigational Site, Kingwood, Texas
  - GSK Investigational Site, Nacogdoches, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Williston, Vermont
  - GSK Investigational Site, Arlington, Virginia
  - GSK Investigational Site, Ashburn, Virginia
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Christiansburg, Virginia
  - GSK Investigational Site, Danville, Virginia
  - GSK Investigational Site, Falls Church, Virginia
  - GSK Investigational Site, Midlothian, Virginia
  - GSK Investigational Site, Newport News, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Portsmouth, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Suffolk, Virginia
  - GSK Investigational Site, Virginia Beach, Virginia
  - GSK Investigational Site, Bellingham, Washington
  - GSK Investigational Site, Everett, Washington
  - GSK Investigational Site, Renton, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Charleston, West Virginia
  - GSK Investigational Site, Weirton, West Virginia
  - GSK Investigational Site, Mequion, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin
  - GSK Investigational Site, Racine, Wisconsin
  - GSK Investigational Site, Waukesha, Wisconsin
  - GSK Investigational Site, Wauwatosa, Wisconsin
  - GSK Investigational Site, West Allis, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: SCA40917 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: SCA40917 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SCA40917 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SCA40917 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: SCA40917 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SCA40917 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register